CLINICAL TRIAL: NCT06708715
Title: Stress Reduction After Use of a Haptic Vibrotactile Trigger Technology Patch: Analysis and Assessment
Acronym: STRAVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SuperPatch Limited LLC (Industry)
Collaborators: Clarity Science LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STRAVA-001
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Stress; Anxiety
Keywords: stress; anxiety; SuperPatch; PEACE Patch; Haptic; Vibrotactile Haptic Technology; VTT
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATMENT (Active Comparator): Subjects will be given a patch that incorporates a vibrotactile haptic technology (VTT) sensory pattern (PEACE Patch)
  Interventions: Device: PEACE Patch
- CONTROL (Sham Comparator): Subjects will be given a sham patch that does not incorporate vibrotactile haptic technology.
  Interventions: Device: Topical Sham Patch

INTERVENTIONS:
Device: PEACE Patch — A topical patch that incorporates a sensory pattern of vibrotactile haptic technology.
  Arms: TREATMENT
Device: Topical Sham Patch — Sham Patch that does not include vibrotactile haptic technology
  Arms: CONTROL

SUMMARY:
The purpose of this research study is to collect subject perceptions or feelings about their treatment. Participation includes a survey from individuals who are receiving a stress or anxiety-relieving topical patch [Super Patch PEACE Patch with Haptic Vibrotactile Trigger Technology (VTT)] and assigned to a Treatment Group or given a Sham patch, assigned to the Control Group, to address symptoms or stress and anxiety symptoms using validated scales [for example, The Perceived Stress Scale (PSS) or Medical Outcomes Study Short Form-20 (SF-20)].

DETAILED DESCRIPTION:
This minimal risk observational study, will evaluate an over the counter (OTC) non-invasive, non- pharmacological patch (Super Patch PEACE Patch; The Super Patch Company Ltd LLC., SRYSTY Holding Co., Toronto, Canada) that is embedded with a proprietary sensory pattern and incorporates haptic vibrotactile trigger technology (VTT) and designed to trigger neural pathways and circuits associated with stress, anxiety, and other cortical networks, with other study participants who receive an 'inactive' (Sham) patch without the embedded VTT technology. The sensory patterns within the active patches are in close symmetry between known EEG patterns and their role in modulating EEG and neuronal circuits within higher brain centers.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 85, inclusive
2. Able to provide written informed consent
3. Have received a PEACE Patch from their treating clinician if in treatment group.
4. Is a patient who has been diagnosed with experienced stress or anxiety related issues.
5. Have received a Sham Patch if assigned tot eh Control Group

Exclusion Criteria:

1. Use of drugs of abuse (illicit or prescription)
2. Pregnancy
3. Existing or planned implantation of Pacemaker or other electrical devices

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and Female
Enrollment: 150 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in patient Perceived Stress Scale (PSS) | From enrollment to end of treatment at 2 weeks
  Changes in patient Perceived Stress Scale (PSS) overall scores among and between the treated group and the control group. The Perceived Stress Scale (PSS) score is calculated by adding the score for all 10 questions, after reversing the scores for Q4, 5, 7 and 8 (0=4, 1=3, 2=2, 3=1, 4=0). Total possible score = 40. PSS categorizes stress levels as either high (scores of between 27-40), moderate (scores between 14-26), or low (scores between 0-14).
Changes in patient Medical Outcomes Study Short Form-20 (SF-20) | From enrollment to end of treatment at 2 weeks
  Changes in patient Medical Outcomes Study Short Form-20 (SF-20) for 6 domains among and between the treated group and the control group. There are 20 items and 6 domains in the SF-20 that are measured. These are Physical Functioning, Role Functioning, Social Functioning, Mental Health, Health Perceptions, and Pain. Except for the Pain domain, the higher the percentage, the better the quality-of-life is corresponding. For the Pain domain, the lower the percentage, the lower the amount of bodily pain is corresponding. For the Mental Health domain, the analysis represents the four major mental health dimensions. These are anxiety, depression, loss of behavioral-emotional control, and psychological well- being.
Changes in the use of prescription and OTC medications | From enrollment to end of treatment at 2 weeks
  Changes in Number of Prescription Medications Used based on subject and clinician reporting through a questionnaire for those subjects in Treatment Arm and receiving the active patch (PEACE) or Control Sham patch during study period. Comparisons will be made between prescription medication usage reporting at baseline, 7-day, and 14 days.
Demographics and patient satisfaction with the PEACE Patch treatment. | From enrollment to end of treatment at 2 weeks
  Demographics and patient satisfaction based on subject and clinician reporting for those subjects in Treatment Arm and receiving the active patch (PEACE) or Control Sham patch during study period.

OTHER OUTCOMES:
Any side effects reported by patients will be documented and assessed by clinician and PI | From enrollment to end of treatment at 2 weeks
  Evaluation of reported side effects during study period based on self-report by subject or reported by clinician investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Gudin, MD, Principal Investigator — University of Miami
Locations (1):
- Stein Medical, Tyrone, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided